CLINICAL TRIAL: NCT00822042
Title: Study of Histological and Adipokines Expression Variations in Lipodystrophic Adipose Tissue During Corticosteroids-induced Lipodystrophy
Brief Title: Corticosteroid-induced Lipodystrophy and Adipokines
Acronym: ADIPOKINES
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P 051037; CIRC 05147
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2009-01

CONDITIONS: Lipodystrophy
Keywords: Lipodystrophy; Adipokines; Glucocorticoids; Patients with glucocorticoids
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cytopunction (adipocytes), whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with corticotherapy lasting more than 3 months
  Interventions: Other: Samples and procedures

INTERVENTIONS:
Other: Samples and procedures — * Scanner, histomorphometry : at the inclusion and M3 visits
  * whole blood samples, cytoponction : at the inclusion and M3 visits

SUMMARY:
Hypothesis: systemic therapy with corticosteroid induces morphological changes (e.g., moon face, buffalo neck) called lipodystrophy (LD). We hypothesize that this LD is associated with variation of adipocytokines (e.g., adiponectin, leptine, IL6) levels

Primary objective: To show a 50% decrease in adipocytes adiponectin's expression in patients who developed LD versus those who did not developed LD during the first 3 months of a systemic therapy with corticosteroids

Secondary objectives: To look for differences in the mRNA expression of 11bHSD1, SREBP1c and PPARg in fat samples of patients before and after treatment with systemic corticosteroids and between LD+ and LD-patients To compare the fat morphology before and after treatment with glucosteroids

DETAILED DESCRIPTION:
Design: Monocentric, cross-sectional analytical study

Subjects: 32 HIV-free and Cushing disease-free adult patients for whom a prolonged treatment (³3months) with glucosteroids (³ 0.5 mg/kg/day) is initiated

Methods: At treatment initiation and 3 months after: comparison of fat sample mRNA expression of adipokines (adiponectin, leptin, IL6, TNFa), 11bHSD1, SREBP1c and PPARg, fat morphology and seric concentrations of adiponectin, leptin, IL6, sTNFR1 between patients LD+ and patients LD-. The diagnosis of LD will be performed by 3 experts using patients photographs

Aims of this study:

* To gain a better understanding of the pathophysiology of glucosteroids-induced LD
* To compare this pathophysiology to the one of HIV-associated LD for which the hypothesis of a local, cellular, hypercorticism has been put forward and for which related treatment have been prescribed.

ELIGIBILITY:
Inclusion Criteria:

* adult patient
* starting therapy with prednisone
* corticosteroid therapy lasting more than 3 months
* baseline prednisone dosage >= 0.5 mg/kg/d

Exclusion Criteria:

* Cushing disease
* HIV +Pregnancy
* Recent weight lost (> 5% of the usual weight)
* Therapy with glucocorticosteroids during the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting in participating units
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2006-08; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Expression of adiponectin in adipocytes | at the inclusion and M3 visits

SECONDARY OUTCOMES:
Plasma levels of adiponectin, leptin, sTNFR1, and IL6 | at the inclusion and M3 visits
Histological morphology of adipocytes | at the inclusion and M3 visits
Expression of leptin, IL6, TNFa, 11bHSD1, SREBP1c and PPARg in adipocytes | at the inclusion and M3 visits

CONTACTS AND LOCATIONS:
Overall Officials: Laurence FARDET, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Saint-Antoine, Paris, France